CLINICAL TRIAL: NCT06060301
Title: Adjunctive Effect of Topical Sulfasalazine for Oral Lichen Planus Management: A Randomized Clinical Trial
Brief Title: Topical Sulfasalazine and Oral Lichen Planus
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Zakaria Ibrahium Mohammed, Associate professor Oral Medicine & Periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Faculty of Dentistry, Cairo
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Oral Lichen Planus; Topical Sulfasalazine; Corticosteroids
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Sulfasalazine; Adrenal Cortex Hormones; Orabase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- study group (S group) (Experimental): The patients will use topical sulfasalazine prepared by dissolving one tablet of commercially available in 100 ml of distilled water 4 times per day as a mouth wash combined with topical corticosteroids 4 times per day as a topical gel in an alternate sequence.
  Interventions: Drug: sulfasalazine 500 MG; Drug: corticosteroids
- Control group (C group) (Active Comparator): The 23 patients categorized as control group (C group) will receive topical corticosteroids gel only 4 times per day. The treatment regimen will be continued for 4 weeks.
  Interventions: Drug: corticosteroids

INTERVENTIONS:
Drug: sulfasalazine 500 MG — The patients will use topical corticosteroids in addition to topical sulfasalazine 4 times per day.
  Other Names: colosalazine
  Arms: study group (S group)
Drug: corticosteroids — The patients will use topical corticosteroids 4 times per day.
  Other Names: kenakort in orabase

SUMMARY:
Oral lichen planus (OLP) is a chronic inﬂammatory disease that affects the mucosal membrane. T-cell mediated damage against the mucosal epithelial cells is implicated in the pathogenesis of OLP, although the exact mechanism is unknown.

Sulfasalazine is extensively used in inﬂammatory bowel disease and is effective on immune-related inﬂammatory disease such as Crohn's disease, rheumatoid arthritis, and Behcet's disease. In spite of its effectiveness, the anti-inﬂammatory mechanism is not clearly understood.

DETAILED DESCRIPTION:
* Patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University.
* A total number of 46 patients will be included in this study. The 23 patients categorized as study group (S group) will use topical sulfasalazine prepared by dissolving one tablet of commercially available (COLOSALAZINE - EC 500 MG 20 TAB, manufactured by: Alexandria Company for Pharmaceuticals & Chemical Industries, Alexandria) in 100 ml of distilled water 4 times per day as a mouth wash combined with topical corticosteroids 4 times per day as a topical gel in an alternate sequence. There are no expected side effects of this treatment due to its topical application however, the patient will be instructed to stop the treatment if any adverse reactions occur such as allergy and coming to the clinic next day.
* The 23 patients categorized as control group (C group) will receive topical corticosteroids gel only 4 times per day. The treatment regimen will be continued for 4 weeks with follow up visits one per week.
* Medical history will be taken, thorough oral examination will be done, and a full questionnaire will be filled for each patient.
* All participants in the study groups will undergo adequate oral hygiene performance measures with complete removal of plaque and calculus as they implement intraoral inflammation and intensify both extension and symptoms of OLP lesions. Patients will be advised to evade accidental trauma on soft tissues using soft bristles toothbrush. Acidic, spicy, hard, hot food and beverages will be avoided.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with 30-65 years old
* Patents with atrophic OLP

Exclusion Criteria:

* - Smokers
* pregnant or lactating ladies and
* Patients under topical or systemic steroids during the last two months
* Patients using lichenoid reaction-inducing drugs,
* Patients with positive hepatitis C virus (HCV) antibodies, diabetes and hypertension
* Patients having amalgam filling adjacent lesions will not also be included

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
NAS | Every week for 4 weeks period
  Scale for pain assessment
sign scoring scale of Thongprasom | Every week for 4 weeks period
  Score for severity

CONTACTS AND LOCATIONS:
Overall Officials: Faculty O Dentistry, Cairo University, Study Chair — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Because the research not published yet.